CLINICAL TRIAL: NCT02925702
Title: Prospective Multi-centre Study of Prognostic Factors in Metastatic Castration-Resitant Prostate Cancer Patients Treated With Radium-223.
Brief Title: PRORADIUM: Prospective Multi-centre Study of Prognostic Factors in mCRPC Patients Treated With Radium-223.
Acronym: PRORADIUM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centro Nacional de Investigaciones Oncologicas CARLOS III (Other)
Collaborators: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Other Study IDs: IBIMA-CNIO-CP-03-2015; CNI-RAD-2016-01 (Other: CNIO)
Record Dates: First submitted 2016-09-29; First posted 2016-10-06 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2019-02

CONDITIONS: Advanced Prostate Cancer; Castration Resistant; Radium 223
Keywords: metastatic Castration Resistant Prostate Cancer; Radium-223; Biomarkers
MeSH Terms: interventions — radium Ra 223 dichloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and FFPE
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Radium-223: Radium-223 55 mBq/Kg every 4 weeks IV
  Interventions: Drug: Radium 223 55mBq/Kg every 4 weeks intravenously

INTERVENTIONS:
Drug: Radium 223 55mBq/Kg every 4 weeks intravenously — Radium-223 55kBq/kg infusion IV every 4 weeks
  Other Names: radium-223 dichloride; Xofigo®

SUMMARY:
PRORADIUM is a prospective multicentre observational study in metastatic Castration-Resistant Prostate Cancer (mCRPC), designed to explore prognostic biomarkers in patients undergoing treatment with radium-223.

DETAILED DESCRIPTION:
This study is a prospective biomarker study of patients with mCRPC undergoing treatment with radium-223 as standard of care treatment. The participants will undergo serial pre- and post-therapy blood collection for biomarker analysis as part of the primary objective of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male age ≥ 18 years
2. Histologically confirmed adenocarcinome of the prostate
3. ECOG Performance Status ≤ 2
4. Castration resistance must be documented with surgical or medical castration with serum testosterone < 50 ng/mL (< 2.0 nM).
5. Men diagnosed with at least one metastatic lesion on CT or bone scan.
6. Documented biochemical and/or radiographic progression to previous treatment according to PCWG2 criteria.
7. Patients who are candidates for standard of care treatment with Radium-223 55mBq/Kg very 4 weeks intravenously
8. Availability of formalin-fixed paraffin-embedded blocks from the prostate biopsy and/or radical prostatectomy.
9. Acceptable hematological, hepatic and renal functions.

Exclusion Criteria:

1. Previous cancer diagnosis, except those patients who had a localized malignant tumour and who are five years cancer-free or those diagnosed with skin cancers (of non-melanoma type) or excised in situ carcinomas.
2. Any condition or reason that, in the opinion of the Investigator, interferes with the ability of the patient to participate in the trial, which places the patient at undue risk, or complicates the interpretation of safety data

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: metastatic Castration-Resistant Prostate Cancer
Sampling Method: Non-Probability Sample
Enrollment: 161 (Estimated)
Dates: Start 2016-02; Primary Completion 2019-01 (Actual); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
To validate the prognostic value for overall survival of serum bone metabolism markers descibed by Primo N Lara et al (JNCI 2014) in mCRPC patients treated with Radium-223 | Initially 48 months, currently 60 months

SECONDARY OUTCOMES:
To analyze the prognostic value for biochemical and/or radiological progression-free survival of serum bone metabolism markers described by Primo N Lara et al in mCRPC patients treated with Radium-223 | Initially 48 months, currently 60 months
To assess the prognostic value of alkaline phosphatase before- and after 3 cycles of treatment in these patients | Initially 48 months, currently 60 months
To analyze the prognostic value of "Bone Scan Index" in mCRPC patients treated with Radium-223 | Initially 48 months, currently 60 months
To assess the prognostic value for overall survival of androgen receptor splicing variant 7 (AR-V7) and/or AR amplification in mCRPC patients treated with Radium-223 | Initially 48 months, currently 60 months
To validate the prognostic value of the gene-expression signature from peripheral blood described by Olmos et al (Lancet Oncol 2012) on overall survival of mCRPC patients | Initially 48 months, currently 60 months
To correlate the presence of somatic and/or germinal mutations with the outcomes of these patients | Initially 48 months, currently 60 months
Exploratory aims include: Validate the prognostic value of classical nomograms designed to assess the outcomes of mCRPC patients and analyze the prognostic value of the gene-expression signature described by Olmos et al on progression-free survival. | Initially 48 months, currently 60 months

CONTACTS AND LOCATIONS:
Overall Officials: David Olmos, MD, Study Chair — CNIO-Centro Nacionald e Investigaciones Oncológicas; Elena Castro, MD, Study Chair — CNIO-Centro Nacionald e Investigaciones Oncológicas; Rafael Morales, MD, Study Chair — Hospital Vall d'Hebron; Maria Isabel Saez, MD, Study Chair — Hospital Universitario Virgen de la Victoria
Locations (63):
- Spain (63):
  - Hospital Arquitecto Marcide, Ferrol, A Coruña
  - Hospital Universitario de Santiago, Santiago de Compostela, A Coruña
  - Hospital Universitario de Elche, Elche, Alicante
  - Hospital San Llatzer, Palma de Mallorca, Balearic Islands
  - ICO L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Althaia Manresa, Manresa, Barcelona
  - Hospital de Mataró, Mataró, Barcelona
  - Hospital Parc Taulí, Sabadell, Barcelona
  - Hospital Moisès Broggi, Sant Joan Despí, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Hospital Marqués de Valdecilla, Santander, Cantabria
  - Hospital de Especialidades de Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - Hospital Onkologikoa, Instituto Oncológico de Kutxa, Donostia / San Sebastian, Guipúzcoa
  - Hospital San Pedro de La Rioja, Logroño, La Rioja
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas, Las Palmas de Gran Canaria
  - Fundación Hospital de Alcorcón, Alcorcón, Madrid
  - Hospital Universitario Quirón, Pozuelo de Alarcón, Madrid
  - Hospital Infanta Sofía, San Sebastián de los Reyes, Madrid
  - Hospital Costa del Sol, Marbella, Málaga
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Complejo Hospitalario Universitario de Vigo, Vigo, Pontevedra
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital Lluis Alcanyis, Xátiva, Valencia
  - Fundacion Centro Oncologico de Galicia, A Coruña
  - Hospital Nuestra Señora de Sonsoles, Ávila
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall D'Hebron, Barcelona
  - Nuclear Medicine Coordination PROCURE-PRORADIUM, Barcelona
  - Hospital de Burgos, Burgos
  - Hospital Puerta del Mar, Cadiz
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital de Ciudad Real, Ciudad Real
  - Hospital Universitario Reina Sofia, Córdoba
  - Instituto Catalán de Oncología de Girona-ICO Girona, Girona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario de Guadalajara, Guadalajara
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Lucus Augusti, Lugo
  - Hospital Universitario Gregorio Maranon, Madrid
  - CNIO-Centro Nacional de Investigaciones Oncológicas, Madrid
  - Coordination PROCURE-Centro Nacional de Investigaciones Oncologicas, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Centro Integral Oncologico Clara Campal, Madrid
  - Anatomical Pathology PROCURE, Málaga
  - Hospital Regional Universitario Virgen de la Victoria, Málaga
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Morales Messeguer, Murcia
  - Complejo Hospitalario Universitario de Ourense, Ourense
  - Hospital Son Espases, Palma de Mallorca
  - Complejo Hospitalario de Pontevedra, Pontevedra
  - Hospital Clínico de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universxitario Nuestra Señora de Valme, Seville
  - Hospital Virgen de la Salud-Complejo Hospitalario de Toledo, Toledo
  - Fundación Instituto Valenciano de Oncología, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Arnau Vilanova, Valencia
  - Hospital Universitario La Fe, Valencia
  - Hospital Clínico Lozano Blesa, Zaragoza

REFERENCES:
- [Derived] Romero-Laorden N, Lorente D, de Velasco G, Lozano R, Herrera B, Puente J, Lopez PP, Medina A, Almagro E, Gonzalez-Billalabeitia E, Villla-Guzman JC, Gonzalez-Del-Alba A, Borrega P, Lainez N, Fernandez-Freire A, Hernandez A, Rodriguez-Vida A, Chirivella I, Fernandez-Parra E, Lopez-Campos F, Isabel Pacheco M, Morales-Barrera R, Fernandez O, Villatoro R, Luque R, Hernando S, Castellano DC, Castro E, Olmos D. Prospective Assessment of Bone Metabolism Biomarkers and Survival in Metastatic Castration-resistant Prostate Cancer Patients Treated with Radium-223: The PRORADIUM Study. Eur Urol Oncol. 2024 Jun;7(3):447-455. doi: 10.1016/j.euo.2023.09.015. Epub 2023 Oct 12. PMID 37838555